CLINICAL TRIAL: NCT04140825
Title: Within-Breath Total Respiratory Input Impedance in Healthy Adult Subjects
Status: Completed | Type: Observational
Sponsor: Restech Srl (Industry)
Collaborators: MGC Diagnostics (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1/17 ADU
Record Dates: First submitted 2019-06-27; First posted 2019-10-28 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Respiratory Disease
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Group 1: Subjects>=18 years old will measure as a minimum FOT and spirometry.
  Interventions: Device: Resmon PRO FULL

INTERVENTIONS:
Device: Resmon PRO FULL — Measurement of lung impedance by the Forced Oscillation Technique

SUMMARY:
Assessment of lung function requires the evaluation of pulmonary function by spirometry. However, some patients (e.g. children, elderly, or diseased individuals) may have difficulty performing the related forced maximal respiratory maneuver correctly. Forced oscillation technique (FOT) is increasingly being used in clinical settings to evaluate lung function noninvasively by measuring the mechanical input impedance of the respiratory system. FOT measures lung impedance during tidal breathing, requiring minimal patient cooperation. Recently a new methodology (within breath analysis) has emerged to evaluate changes that occur in the impedance during the breathing activity. The within-breath calculation of impedance allows separating the contribution of inspiration and expiration to the measured parameters.

The purpose of this study is to establish reference ranges for within breath FOT parameters and their short term variability.

DETAILED DESCRIPTION:
Purpose and rationale Assessment of lung function requires the evaluation of pulmonary function by spirometry. However, some patients (e.g. children, elderly, or diseased individuals) may have difficulty performing the related forced maximal respiratory maneuver correctly. Forced oscillation technique (FOT) is increasingly being used in clinical settings to evaluate lung function noninvasively by measuring the mechanical input impedance of the respiratory system. FOT measures lung impedance during tidal breathing, requiring minimal patient cooperation. Recently a new methodology (within breath analysis) has emerged to evaluate changes that occur in the impedance during the breathing activity. The within-breath calculation of impedance allows separating the contribution of inspiration and expiration to the measured parameters.

The purpose of this study is to establish reference ranges for within breath FOT parameters and their short term variability.

Objectives Primary: To derive equations to predict normal values and normality ranges for within-breath respiratory system resistance, reactance and related parameters at the selected stimulating waveform and to measure the short term variability of such parameters.

Secondary: To demonstrate the equivalence of the results of a single multiple-breath test to results obtained as an average of 3 consecutive repeated tests.

Study design This will be a prospective multi-center trial of healthy subjects. After signing the Informed Consent, an interview and physical examination will be performed. The examiner will confirm that subjects are able to perform acceptable and repeatable spirometry. FOT measurements will be performed, followed by standard spirometry measurements.

Study Duration This is a single visit study. Subject participation will be completed in 1 hour and 15 min. Enrollment of all subjects is expected to take 23 weeks (6 months).

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years of age.
* Signature of the written informed consent

Exclusion Criteria:

Subjects will be excluded if they meet at least one of the following conditions:

* Abnormal spirometry defined as FEV1, FEV1/VC and VC below the LLN as established by the Global Lung function (GLI) 2012 reference equations.
* Smokers or ex-smokers
* BMI >30 kg/cm2
* History of respiratory symptoms using the ECRHS II screening questionnaire (www.ecrhs.org)

  * Wheezing
  * Cough
  * Phlegm production
  * Dyspnea
  * Feeling of chest tightness
  * Night awakening due to a cough attack
* Have a history of pulmonary or cardiac disease
* Had a recent (e.g., in the last 4 weeks) respiratory tract infection
* Have a neurological or neuromuscular disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The following group will be considered:
  Adults (>= 18 years old)
Sampling Method: Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Correlation between respiratory impedance parameters and the following variables: age, height, weight, sex, abdominal circumference and phenotype, breathing pattern parameters. | 1 day
  The equation resulting from the multivariate regression analysis between impedance parameters assessed during the test and anthropometric measurements of age, height, weight, sex, abdominal circumference and phenotype, breathing pattern parameters

SECONDARY OUTCOMES:
Noninferiority of one FOT test vs. the average of three consecutive tests | 1 day
  Noninferiority hypothesis of the results of a single test with multiple breaths free from artifacts compared to those obtained in the same session as an average or 3 consecutive repeated tests

CONTACTS AND LOCATIONS:
Overall Officials: David Kaminsky, MD, Principal Investigator — University of Vermont Medical Center Inc
Locations (4):
- United States (2):
  - Biomedical Research Institute at Harbor- UCLA Medical Center, Los Angeles, California
  - University of Vermont Medical Center Inc., Burlington, Vermont
- Italy (2):
  - Catholic University of the Sacred Heart, Rome, RM
  - U.O.C. Malattie dell'apparato respiratorio e endoscopia delle vie aeree - Ospedale San Giovanni, Roma, Rome

REFERENCES:
- [Background] DUBOIS AB, BRODY AW, LEWIS DH, BURGESS BF Jr. Oscillation mechanics of lungs and chest in man. J Appl Physiol. 1956 May;8(6):587-94. doi: 10.1152/jappl.1956.8.6.587. No abstract available. PMID 13331841
- [Background] Peslin R, Ying Y, Gallina C, Duvivier C. Within-breath variations of forced oscillation resistance in healthy subjects. Eur Respir J. 1992 Jan;5(1):86-92. PMID 1577156
- [Background] Horowitz JG, Siegel SD, Primiano FP Jr, Chester EH. Computation of respiratory impedance from forced sinusoidal oscillations during breathing. Comput Biomed Res. 1983 Dec;16(6):499-521. doi: 10.1016/0010-4809(83)90037-x. PMID 6653086
- [Background] Dellaca RL, Santus P, Aliverti A, Stevenson N, Centanni S, Macklem PT, Pedotti A, Calverley PM. Detection of expiratory flow limitation in COPD using the forced oscillation technique. Eur Respir J. 2004 Feb;23(2):232-40. doi: 10.1183/09031936.04.00046804. PMID 14979497
- [Background] Dellaca RL, Pompilio PP, Walker PP, Duffy N, Pedotti A, Calverley PM. Effect of bronchodilation on expiratory flow limitation and resting lung mechanics in COPD. Eur Respir J. 2009 Jun;33(6):1329-37. doi: 10.1183/09031936.00139608. Epub 2009 Jan 22. PMID 19164347
- [Background] Pasker HG, Schepers R, Clement J, Van de Woestijne KP. Total respiratory impedance measured by means of the forced oscillation technique in subjects with and without respiratory complaints. Eur Respir J. 1996 Jan;9(1):131-9. doi: 10.1183/09031936.96.09010132. PMID 8834346
- [Background] Brown NJ, Xuan W, Salome CM, Berend N, Hunter ML, Musk AW, James AL, King GG. Reference equations for respiratory system resistance and reactance in adults. Respir Physiol Neurobiol. 2010 Jul 31;172(3):162-8. doi: 10.1016/j.resp.2010.05.013. Epub 2010 May 15. PMID 20478414
- [Background] Aarli BB, Eagan TM, Ellingsen I, Bakke PS, Hardie JA. Reference values for within-breath pulmonary impedance parameters in asymptomatic elderly. Clin Respir J. 2013 Jul;7(3):245-52. doi: 10.1111/j.1752-699X.2012.00312.x. Epub 2012 Aug 20. PMID 22822726
- [Background] Oostveen E, MacLeod D, Lorino H, Farre R, Hantos Z, Desager K, Marchal F; ERS Task Force on Respiratory Impedance Measurements. The forced oscillation technique in clinical practice: methodology, recommendations and future developments. Eur Respir J. 2003 Dec;22(6):1026-41. doi: 10.1183/09031936.03.00089403. PMID 14680096
- [Background] Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall GL, Culver BH, Enright PL, Hankinson JL, Ip MS, Zheng J, Stocks J; ERS Global Lung Function Initiative. Multi-ethnic reference values for spirometry for the 3-95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012 Dec;40(6):1324-43. doi: 10.1183/09031936.00080312. Epub 2012 Jun 27. PMID 22743675
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Wanger J, Clausen JL, Coates A, Pedersen OF, Brusasco V, Burgos F, Casaburi R, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson D, Macintyre N, McKay R, Miller MR, Navajas D, Pellegrino R, Viegi G. Standardisation of the measurement of lung volumes. Eur Respir J. 2005 Sep;26(3):511-22. doi: 10.1183/09031936.05.00035005. No abstract available. PMID 16135736
- [Background] Calogero C, Simpson SJ, Lombardi E, Parri N, Cuomo B, Palumbo M, de Martino M, Shackleton C, Verheggen M, Gavidia T, Franklin PJ, Kusel MM, Park J, Sly PD, Hall GL. Respiratory impedance and bronchodilator responsiveness in healthy children aged 2-13 years. Pediatr Pulmonol. 2013 Jul;48(7):707-15. doi: 10.1002/ppul.22699. Epub 2012 Nov 20. PMID 23169525
- [Background] Ducharme FM, Davis GM, Ducharme GR. Pediatric reference values for respiratory resistance measured by forced oscillation. Chest. 1998 May;113(5):1322-8. doi: 10.1378/chest.113.5.1322. PMID 9596314
- [Background] Oostveen E, Boda K, van der Grinten CP, James AL, Young S, Nieland H, Hantos Z. Respiratory impedance in healthy subjects: baseline values and bronchodilator response. Eur Respir J. 2013 Dec;42(6):1513-23. doi: 10.1183/09031936.00126212. Epub 2013 Apr 18. PMID 23598954
- [Background] Knofczynski, G. T. & Mundfrom, D. Sample Sizes When Using Multiple Linear Regression for Prediction. Educ. Psychol. Meas. 68, 431-442 (2007).